CLINICAL TRIAL: NCT02797236
Title: A Phase I Dose Escalation Study to Assess the Safety and Immunogenicity of the SF2a-TT15 Conjugate Vaccine Against S. Flexneri 2a in Healthy Adult Volunteers
Brief Title: SF2a-TT15 Conjugate Vaccine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-060
Record Dates: First submitted 2016-04-18; First posted 2016-06-13 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Shigellosis; Bacillary Dysentery
Keywords: Phase I; conjugate vaccine; Shigella flexneri 2a; safety; Immunogenicity; Healthy adults
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- vaccine dose 1 (Experimental): SF2a-TT15 vaccine, 2 μg
  Interventions: Biological: SF2a-TT15 vaccine
- vaccine dose 1+ adjuvant (Experimental): SF2a-TT15 vaccine, 2 μg + alum
  Interventions: Biological: SF2a-TT15 vaccine + adjuvant
- vaccine dose 2 (Experimental): SF2a-TT15 vaccine, 10 μg
  Interventions: Biological: SF2a-TT15 vaccine
- vaccine dose 2 + adjuvant (Experimental): SF2a-TT15 vaccine, 10 μg + alum
  Interventions: Biological: SF2a-TT15 vaccine + adjuvant
- Placebo (Placebo Comparator): Tris buffer
  Interventions: Biological: Placebo
- Placebo + adjuvant (Placebo Comparator): Tris buffer + Alum
  Interventions: Biological: Placebo + adjuvant

INTERVENTIONS:
Biological: SF2a-TT15 vaccine
  Arms: vaccine dose 1; vaccine dose 2
Biological: SF2a-TT15 vaccine + adjuvant
  Arms: vaccine dose 1+ adjuvant; vaccine dose 2 + adjuvant
Biological: Placebo
  Arms: Placebo
Biological: Placebo + adjuvant
  Arms: Placebo + adjuvant

SUMMARY:
This is a first-in-human, single-center, single-blinded, observer-masked randomized, dose escalation (two doses), placebo-controlled study in healthy volunteers.

DETAILED DESCRIPTION:
Subjects will be assigned to one of two cohorts.

1. Cohort 1 will receive the lower dose of 2 μg vaccine (with or without alum adjuvant) or matching placebo.
2. Cohort 2 will receive the higher dose of 10 μg vaccine (with or without alum adjuvant) or matching placebo.

Eligible subjects will be randomized to receive the 2 μg dose or 10 µg without or with alum or matching placebo, at a ratio of 3:1, as three single IM injections. There will be an interval of 28(±3) days) between each treatment.

The study will be conducted in a stepwise approach in which a "Pioneer" Group of 2 subjects (one receiving the active vaccine and one receiving the matching placebo) will receive the first injection. These subjects will remain in-house for a 24-hours medical observation after the first injection (not required in the subsequent injections) Once it has been established that there are no safety concerns in the non-adjuvanted "Pioneer" Groups (and after no less than 48 hrs), the next "Pioneer" group (one subject receiving adjuvanted 2 μg vaccine and one receiving the matching alum placebo) will be injected.

If no safety concerns are raised in this group also, after no less than 48 hrs, the rest of the subjects may receive the first injection.

ELIGIBILITY:
Inclusion criteria

* Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
* Negative human leukocyte antigen (HLA) -B27 and no history of reactive arthritis
* Negative HIV, Hepatitis B and Hepatitis C serology tests.
* Blood levels of Shigella flexneri 2a LPS IgG antibodies ≤ percentile 80
* No known history of alcohol abuse

Exclusion criteria

* Subjects with a history of clinically significant gastrointestinal disorders or with any history of frequent diarrhea, nausea or emesis, regardless of etiology.
* Individuals with immunosuppressive diseases or under immunosuppressive therapy
* History of culture-proven S. flexneri.
* Individuals who have household contact with/and /or intimate exposure to an individual with laboratory confirmed S. flexneri.
* Having travelled in countries/areas highly endemic for S. flexneri within 3 months prior to enrolment.
* Previous participation in any study in which a Shigella-vaccine candidate was administered.
* Known contraindication, hypersensitivity and/or allergy to the investigational product or its excipients.
* Known hypersensitivity and/or allergy to any drug or vaccine
* Women who are pregnant or are breast-feeding, or are of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 12 months
  Safety: Occurrence, frequency, severity, and duration of local and systemic adverse events (AEs) including clinically significant laboratory abnormalities, after administration of the SF2a-TT15 vaccine.

SECONDARY OUTCOMES:
Immunogenicity - humoral Immune response | 12 months
  Serum antibody response (IgG IgM, IgA) to S. flexneri 2a LPS, following the administration of the various vaccine doses and antibody secreting cells to S. flexneri 2a LPS, following the administration of the various vaccine doses

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Souraski Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Cohen D, Atsmon J, Artaud C, Meron-Sudai S, Gougeon ML, Bialik A, Goren S, Asato V, Ariel-Cohen O, Reizis A, Dorman A, Hoitink CWG, Westdijk J, Ashkenazi S, Sansonetti P, Mulard LA, Phalipon A. Safety and immunogenicity of a synthetic carbohydrate conjugate vaccine against Shigella flexneri 2a in healthy adult volunteers: a phase 1, dose-escalating, single-blind, randomised, placebo-controlled study. Lancet Infect Dis. 2021 Apr;21(4):546-558. doi: 10.1016/S1473-3099(20)30488-6. Epub 2020 Nov 10. PMID 33186516